CLINICAL TRIAL: NCT00073632
Title: Developing a New Therapy for GAD: Acceptance-Based CBT
Brief Title: Acceptance-Based Treatment for Generalized Anxiety Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Lizabeth Roemer, Ph. D., University of Massachusetts Boston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21MH063208 (NIH); R21MH063208 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-12-02; First posted 2003-12-03 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2008-09

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Acceptance Based Behavioral Therapy

SUMMARY:
This study will develop and implement an awareness- and acceptance-based for treatment of individuals with generalized anxiety disorder.

DETAILED DESCRIPTION:
Participants in this study are recruited from intakes at the Center for Anxiety and Related Disorders at Boston University. Participants will be randomly assigned to receive either acceptance and mindfulness-based strategies plus cognitive behavioral therapy or no treatment for 16 weeks. The treatment will involve daily practice of mindfulness techniques to help draw attention to and accept various emotional states. Interviews, questionnaires, and depression and anxiety scales will be used to assess participants. Assessments will be conducted post-treatment and at 3- and 9-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Generalized Anxiety Disorder (GAD)
* Willing to maintain medication levels and refrain from any additional psychosocial treatment during the course of the study

Exclusion Criteria:

* Bipolar disorder, psychotic disorder, or substance dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-05; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Clinician Severity Rating from ADIS for GAD | pre, post, 3 mo. f/u, 9 mo. f/u
Penn State Worry Questionnaire | pre-, post-, 3 mo. f/u, 9 mo. f/u
Depression Anxiety and Stress Scales, anxiety and stress subscales | pre-, post-, 3 mo. f/u, 9 mo. f/u

CONTACTS AND LOCATIONS:
Overall Officials: Lizabeth Roemer, PhD, Principal Investigator — University of Massachusetts, Boston; Susan M Orsillo, PhD, Principal Investigator — Boston University
Locations (1):
- Center for Anxiety and Related Disorders, Boston, Massachusetts, United States

REFERENCES:
- [Background] Roemer L, Orsillo SM. An open trial of an acceptance-based behavior therapy for generalized anxiety disorder. Behav Ther. 2007 Mar;38(1):72-85. doi: 10.1016/j.beth.2006.04.004. Epub 2006 Oct 24. PMID 17292696